CLINICAL TRIAL: NCT05999903
Title: Driving Rehabilitation and Innovation for Evaluating Risk in Post-Intensive Care Unit Survivors
Acronym: DRIVE-PICS
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Wisconsin, Madison (Other); University of Texas at Austin (Other); Vanderbilt University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R21AG080339-01 (NIH); 1R21AG080339-01 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Delirium; Critical Illness; Drive
Keywords: Adult; Human; Vehicle Driving; Functional Outcomes; Post-Intensive Care Syndrome (PICS); Neuro-Psychological; Cognitive; Neuro Cognitive; Intensive Care Unit (ICU); Longitudinal
MeSH Terms: conditions — Delirium; Critical Illness; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Kinematic Driving Data: Longitudinal kinematic driving data paired with neurocognitive assessments at 3- and 6-months

SUMMARY:
Older adults are at risk for ICU-acquired cognitive decline discernible from clinical, biological, and imaging- related changes in the brain following delirium and critical illness. Our Driving Rehabilitation and Innovation for Evaluating Risk in Post Intensive Care Unit Survivors (DRIVE-PICS) application seeks to implement in-vehicle kinematic driving data with neurocognitive assessments for essential formative work to develop data-based insights into driving behaviors. DRIVE-PICS is designed to contribute to a critical gap in health promotion to develop an evidence-based, in-vehicle driving assessment system to provide actionable driving safety data and rehabilitation strategies tailored to older ICU survivors, the participants' care partners, and clinicians.

DETAILED DESCRIPTION:
There are more than 50 million older adults licensed to drive in the United States. Driving is a complex task requiring cognitive and sensorimotor skills. Survivors of critical illness experience cognitive, psychological and physical impairments, known as Post-Intensive Care Syndrome (PICS), that can last months to years following critical illness. Across the lifespan, ICU recovery has far-reaching implications for independent functioning, employment, and healthcare utilization, costing billions annually. Older adults are at risk for ICU- acquired cognitive decline discernible from clinical, biological, and imaging-related changes in the brain following delirium and critical illness. Similar to other forms of dementia, the combination of normal aging paired with cognitive deficits associated with critical illness survivorship places these older adults at high risk of automobile crashes. To address ICU-acquired cognitive decline, driving assessments to characterize risky driving behaviors are promising to guide driving rehabilitation and intervention development. Rigorous and reproducible driving safety assessment programs have demonstrated success in post-stroke and dementia contexts, established via in-vehicle and virtual modes. The investigators hypothesize that in-vehicle driving assessment and monitoring is a feasible and acceptable approach to assess and address ICU survivor driving safety. The investigators seek to implement novel in-vehicle cloud-data collection technology developed by the investigators' team. The investigators propose to pair neurocognitive assessments with in-vehicle kinematic driving data to conduct essential formative work to develop data-based insights into driving behaviors of older adults with ICU-acquired cognitive declines. The investigators aim to determine protocol feasibility and acceptability of neurocognitive assessments and in-vehicle sensor deployment (Aim 1). The investigators will enroll a cohort of older ICU survivors (n=24) with risk factors for ICU-acquired cognitive impairment to complete neurocognitive measures and participate in driving data collection via in-vehicle sensors over a 6-month post-hospital discharge period. Next, the investigators will evaluate the relationship between neurocognitive assessments and driving behavior and safety in older ICU survivors (Aim 2). Lastly, the investigators will conduct stakeholder advisory panels on the priorities and data presentation needs of driving assessments for older ICU survivors (Aim 3). The stakeholder advisory panel insights will provide scientific justification and protocol feasibility to evaluate recruitment, acceptability and attrition for future full-scale implementation. As the population of older drivers grows, almost doubling in size from 2012 to 2040 there is an immediate and critical need to address this impactful issue. This work is designed in response to the NIA Strategic Plan (Goal C-1-9 Safety of Older Drivers) to contribute to a critical gap in health promotion to develop an evidence-based, in- vehicle driving assessment system to provide actionable driving safety data and rehabilitation strategies tailored to ICU survivors, the participants' care partners and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 and older.
* Must have had an ICU stay with delirium.
* Expected to survive hospital discharge.
* English proficiency
* Active driver within 4 weeks prior to index hospitalization
* Regular use of vehicle that is model year 1996 or newer

Exclusion Criteria:

* Communication challenges due to severe pre-existing dementia, hearing, or vision impairment.
* No access to driving.
* Loss or suspension of driver's license
* Current Incarceration

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU survivors
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Total Driving Time | 0-6 months after hospital discharge
  Total driving time in minutes.

SECONDARY OUTCOMES:
Depression | Hospital discharge, 3 months after hospital discharge, 6 months after hospital discharge
  Depression will be measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report of depression symptoms. Participants rate each item from 0 (not at all) to 3 (very often) to indicate the degree to which they have experienced the symptom in the past 7 days. Higher scores indicate greater depression.
Executive Function | 3 months after hospital discharge, 6 months after hospital discharge
  Executive Function will be measured using the Dimensional Change Card Sort. The participant will be required to sort first according to one dimension (e.g., color) and then according to another dimension (e.g., shape).
Attention | 3 months after hospital discharge, 6 months after hospital discharge
  Attention will be measured using the Flanker Inhibitory Control and Attention Test. The participants will be required to focus on a given stimulus while inhibiting attention to stimuli. Sometimes the middle stimulus points in the same direction as the "flankers" (congruent) and sometimes in the opposite direction (incongruent). if a participant scores ≥ 90%, 20 additional trials with arrows are presented.
Working Memory | 3 months after hospital discharge, 6 months after hospital discharge
  Working memory will be measured using the List Sorting Test. Participants will be provided pictures of different foods and animals accompanied with an audio recording as well as written text. The participant will be asked to recall the items back in size order from smallest to largest, first within a single dimension (either animals or foods, called 1-List) and then on two dimensions (foods, then animals, called 2-List).
Processing Speed | 3 months after hospital discharge, 6 months after hospital discharge
  Processing Speed will be measured using the Pattern Comparison Processing Speed Test. Participants are asked to quickly determine whether two stimuli are the same or not the same. The participants' score will be based on how many items they answer correctly out of a possible 130 items, completed in 90 seconds.
Health-Related Quality of Life | Hospital discharge, 3 months after hospital discharge, 6 months after hospital discharge
  Health-Related Quality of Life will be measured using the EuroQol- 5 Dimension Test (EQ-5D). The participant will be required to answer one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Within the questionnaire, the participants will also be asked to rate their perception of how their health is on a scale of 0 (worst possible health status) to 100 (best possible health status). Questions are scored as a 1 (full health) and 0 (poorest health). With 0 being the worst health status.
Anxiety | Hospital discharge, 3 months after hospital discharge, 6 months after hospital discharge
  Anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report of depression symptoms. Participants rate each item from 0 (not at all) to 3 (very often) to indicate the degree to which they have experienced the symptom in the past 7 days. Higher scores indicate greater depression.
Employment | Hospital discharge, 3 months after hospital discharge, 6 months after hospital discharge
  Employment will be measured through the Johns Hopkins OACIS Employment Questionnaire. It is not a scored questionnaire.
Driving Trips | 0-6 months after hospital discharge
  Driving trips will be measured using the number of trips the participant takes from the beginning of ignition to the end when the vehicle is turned off.
Driving Behaviors | 0-6 months after hospital discharge
  Driving behaviors will be measured using near-crash events that are detected with validated accelerometer thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Danesh, PhD, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor Scott and White Health Medical Center At Temple, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No study documents available.